CLINICAL TRIAL: NCT01452009
Title: Three Month Safety and Efficacy Study of TRAVATAN® vs Travoprost Ophthalmic Solution, 0.004%
Brief Title: Three Month Safety and Efficacy Study of TRAVATAN® Versus Travoprost Ophthalmic Solution, 0.004%
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Management Decision
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-10-151
Record Dates: First submitted 2011-10-12; First posted 2011-10-14 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
Keywords: open angle glaucoma; ocular hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Travoprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Travoprost Ophthalmic Solution, 0.004% (New Formulation) (Experimental)
  Interventions: Drug: Travoprost Ophthalmic Solution, 0.004% (New Formulation)
- TRAVATAN® (Active Comparator): TRAVATAN® administered one drop once daily
  Interventions: Drug: TRAVATAN®

INTERVENTIONS:
Drug: Travoprost Ophthalmic Solution, 0.004% (New Formulation) — Travoprost Ophthalmic Solution, 0.004% given one drop once daily
  Arms: Travoprost Ophthalmic Solution, 0.004% (New Formulation)
Drug: TRAVATAN® — TRAVATAN® administered one drop once daily
  Arms: TRAVATAN®

SUMMARY:
A multi-center, observer-masked, randomized, parallel group efficacy and safety study of TRAVATAN® versus a new formulation of Travoprost Ophthalmic Solution, 0.004%

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older
2. Either gender
3. Any race/ethnicity
4. Diagnosed with open-angle glaucoma (including patients with pseudoexfoliation and pigment dispersion) or ocular hypertension

Exclusion Criteria:

1. Patients with any form of glaucoma other than open-angle glaucoma.
2. Patients with a central cornea thickness greater than 620 μm
3. Patients with Shaffer angle Grade < 2
4. Patients with a cup/disc ratio greater than 0.80
5. Patients with severe central visual field loss
6. Best-Corrected Visual Acuity score worse than 55 ETDRS letters (20/80 Snellen equivalent)
7. Chronic, recurrent or severe inflammatory eye disease
8. Clinically significant or progressive retinal disease
9. Other ocular pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Efficacy: mean IOP Efficacy as measured by mean IOP | 3 months